CLINICAL TRIAL: NCT06543316
Title: Accelerated Marginal Ulcer Healing With Low-Thermal Argon Plasma Endoscopic Treatment
Brief Title: Marginal Ulcer Healing With Low-Thermal Argon Plasma Endoscopic Treatment
Acronym: AMULET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Christopher C. Thompson, MD, MSc (Other)
Collaborators: Erbe USA Incorporated (Other)
Responsible Party: Sponsor-Investigator, Christopher C. Thompson, MD, MSc, Director of Endoscopy, Brigham and Women's Hospital
Organization: Brigham and Women's Hospital (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 2024P002124
Record Dates: First submitted 2024-08-02; First posted 2024-08-09 (Actual); Last update posted 2025-08-05 (Actual); Status verified 2025-07

CONDITIONS: Roux-en-y Anastomosis Site; Marginal Ulcer; Marginal Ulcer (Peptic) or Erosion; Ulcer; Ulcer, Gastric; Ulcer Gastrointestinal; Abdominal Pain; Nausea; Vomiting; GastroIntestinal Bleeding; Dysphagia; Ulcer Gastrojejunal
Keywords: Argon Plasma Coagulation; APC; Low-Thermal Argon Plasma Endoscopic Treatment; Endoscopy; RYGB; Roux-en-Y Gastric Bypass; Ulcer Healing
MeSH Terms: conditions — Peptic Ulcer; Ulcer; Stomach Ulcer; Abdominal Pain; Nausea; Vomiting; Gastrointestinal Hemorrhage; Deglutition Disorders | interventions — Long-Term Potentiation; Therapeutics

STUDY DESIGN:
Intervention Model Description: Randomized, two-arm, crossover clinical study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Low Thermal Plasma (LTP) (Active Comparator): Patients randomized to this group will receive LTP treatment of the ulcer in addition to SOC (PPI administration).
  Interventions: Procedure: Low Thermal Plasma (LTP) Treatment; Other: Standard of Care Ulcer Treatment (typically PPI Administration)
- Standard of Care (SOC) PPI Administration (Active Comparator): Patients randomized to this group will receive only the SOC treatment (PPI administration).
  Interventions: Other: Standard of Care Ulcer Treatment (typically PPI Administration)

INTERVENTIONS:
Procedure: Low Thermal Plasma (LTP) Treatment — For patients randomized to the LTP group, the first LTP treatment will be administered during the initial esophagogastroduodenoscopy (EGD) using a single-use 2.3 mm filtered argon plasma coagulation (FiAPC probe). The argon plasma will be applied at low power settings (~1 W) to the ulcerated areas using pulsed APC effect 0.1.
  Other Names: LTP
  Arms: Low Thermal Plasma (LTP)
Other: Standard of Care Ulcer Treatment (typically PPI Administration) — Standard of care for treatment of ulcers is administration of a proton pump inhibitor (PPI). For patients in the SOC group whose ulcers have not healed completely by the second follow-up at 8 weeks, crossover to LTP treatment will be offered. This treatment will follow the same procedure as the initial LTP treatment.
  Other Names: PPI

SUMMARY:
The objective of the study is to investigate the treatment of marginal ulcers with Low Thermal plasma in an endoscopic setting. By a treatment of the ulcerated areas with argon plasma with low power settings (~ 1 W) we hypothesize that the size of the ulcers will shrink, and the healing is accelerated compared to standard of care alone. Patients will benefit from this minimally invasive approach compared to a much more invasive surgical approach that comes with higher risks and hospital stay length time. From a societal and scientific perspective, this study aims to extend the well-documented clinical benefits of plasma technology - from external wound healing to internal ulcer treatment - within an endoscopic framework. The success of this study could pave the way for broader applications of LTP in the treatment of other endoscopically accessible conditions such as peptic ulcers, duodenal ulcers and esophageal ulcers. This advancement has the potential not only to improve patient outcomes through less invasive methods, but also to position LTP as a cornerstone in the future of gastroenterological wound management strategies.

DETAILED DESCRIPTION:
Gastric bypass surgery, specifically Roux-en-Y gastric bypass (RYGB), is the second most common bariatric procedure performed worldwide (29.3%) after sleeve gastrectomy (55.4%). Despite its success in reducing obesity-related conditions, RYGB is associated with the development of marginal ulcers (MUs)-internal wounds at the gastrojejunal anastomosis prone to poor healing. The incidence of MUs in patients post-RYGB ranges widely, reported at 0.6% to 25% in the U.S., with some estimates as high as 34% worldwide due to asymptomatic cases that go undetected unless investigated endoscopically. These ulcers can become chronic and persisting over time, significantly complicating post-surgical outcomes and increasing the risk of severe complications like perforation, which necessitates urgent surgical intervention in approximately 1-2% of cases.

The current standard of care for MUs involves prolonged use of proton pump inhibitors (PPIs), which reduce gastric acidity to promote ulcer healing. However, this approach addresses only one aspect of MU pathophysiology and is limited by several shortcomings. It is often insufficient in preventing recurrence and carries risks of significant side effects, including increased risk of infection, electrolyte imbalances, and potential kidney disease, particularly with long-term use. Standard therapy is 8 weeks high-dose treatment, and a lifelong PPI therapy is considered if success is seen with medical management. For those not responding to 8 weeks of therapy, most advocate for continued PPI treatment with serial endoscopic evaluation, even up to 2 years out from initial diagnosis. Given these challenges, there is an evident need for alternative treatments that can more effectively target the underlying causes of MUs and reduce the reliance on PPIs.

Low-thermal or low-temperature plasma (LTP) represents a significant advance in accelerated wound healing technologies. As the fourth state of matter, physical plasma is used in the field of plasma medicine to treat a variety of medical conditions at atmospheric pressure and temperatures close to body temperature (typically between 20°C and 50°C). Over the past 10 to 15 years, wound healing has been a primary clinical application for LTP, with extensive use demonstrating its clinical efficacy in the treatment of chronic and poorly healing wounds.

The mechanisms by which LTP facilitates wound healing include oxygenation of tissues, activation of growth factors, improvement of microcirculation, reduction of bacterial load in wounds, and devitalization of senescent cells. These effects are primarily achieved by the ionization of argon gas and the generation of reactive oxygen and nitrogen species (RONS) in the gas phase. Clinically, LTP has been applied to a variety of wound types, including pressure ulcers, chronic wounds, and acute wounds, and has demonstrated effectiveness across a range of wound sizes and stages. LTP treatments are particularly noted for their ability to transform chronic wounds into actively healing wounds, thereby altering the physiological state of the wound.

Several studies have rigorously evaluated the safety profile of LTP and confirmed that it does not pose mutagenic or carcinogenic risks. Long-term evaluations have shown no evidence of tumor formation or abnormal tissue architecture in gas plasma-treated animal models, even after extended periods corresponding to 60 human-equivalent years. Patient follow-up studies using advanced imaging techniques have further confirmed the absence of abnormal healing responses, supporting the absence of adverse long-term effects.

Currently, the most common low-thermal plasma sources used to treat external wounds are PlasmaJets and Dielectric Barrier Discharge (DBD) plasma sources. However, the physical dimensions of these devices limit their use in endoscopic applications. This has limited the availability of LTP for the treatment of internal wounds and ulcers.

Argon plasma coagulation (APC) is a technology that has been used in endoscopy for more than three decades. It has demonstrated clinical safety and efficacy in many areas, including bleeding management (e.g., bleeding ulcers), ablation of cancerous tissue, and precise treatment in sensitive areas. It is primarily used in endoscopic procedures with flexible probes, but also in laparoscopic and open surgery settings. The flexible probes are available in various diameters, 1.5 mm, 2.3 mm and 3.2 mm.

APC works by ionizing argon gas with a high-frequency alternating current passed through an electrode. This ionized gas forms a physical plasma that is applied to tissue. Depending on the mode and effect setting, the plasma can be adjusted in power from as low as 1 W to as high as 120 W. At higher power settings (5 W and above), the plasma exhibits a more pronounced thermal effect due to increased current flow through the tissue, facilitating effective coagulation. Conversely, at lower settings below 5 W, a low-thermal plasma effect is achieved, minimizing tissue coagulation through dynamic application and avoiding prolonged exposure to a single spot. As with PlasmaJets and Dielectric Barrier Discharge (DBD) plasma sources, the effectiveness of low-thermal argon plasma is primarily due to the high energy and voltage that generate reactive oxygen and nitrogen species (RONS).

ELIGIBILITY:
Inclusion Criteria:

* Subjects aged 18 years and above, inclusive of both males and females.
* Patients with a history of Roux-en-Y gastric bypass (RYGB) presenting symptoms indicative of marginal ulcers (MUs) such as abdominal pain, nausea, vomiting, gastrointestinal bleeding, or dysphagia.
* Subjects must be scheduled for an EGD for the evaluation of these symptoms.
* Marginal ulcers confirmed during the initial EGD.
* Willingness to adhere to the SOC treatment, which includes PPIs.
* Subjects able to tolerate repeated endoscopic procedures.
* Capacity for providing informed consent and understanding of study requirements.
* Willingness and ability to attend required follow-up assessments at 4 weeks (+/- 1 week) and 8 weeks (+/- 2 weeks).

Exclusion Criteria:

* Inability to provide informed consent.
* Unwillingness to undergo repeated endoscopies.
* Inability or unwillingness to comply with the SOC.
* Current use of systemic antibiotics.
* Any condition deemed by the investigator to compromise the safety of undergoing an endoscopic procedure.
* Pregnancy, lactation, or absence of reliable contraception in women of childbearing potential.
* Current enrollment in another investigational trial with potential to interfere with this study's endpoint analyses.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-04 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Ulcer Healing Success Rate from baseline endoscopy | Baseline, 4 weeks, 8 Weeks
  Complete healing or significant reduction in ulcer size, determined by endoscopic evaluation at the first follow-up (4 weeks +/- 1 week) and at the end of the second follow-up period (8 weeks +/- 2 weeks).

SECONDARY OUTCOMES:
Comparison of Time to Ulcer Healing between LTP and SOC groups | Baseline, 4 weeks, 8 weeks
  To measure the time in days from initial treatment to complete ulcer healing in both treatment phases, accounting for the initial ulcer size.
Improvement of Tissue Oxygenation at Ulcer Site in LTP treatment group | Baseline, 4 weeks, 8 weeks
  To measure the change of the tissue oxygenation in the ulcerated area directly after the LTP treatment and at the follow-up visits. Level of tissue oxygenation will be compared to a baseline measurement before the initial LTP treatment. Level of tissue oxygenation measured by light absorption with an image sensor (ELUXEO Vision System, Fujifilm).
Presence of Procedure-Related Adverse Events | Baseline, up to 8 weeks
  To evaluate the safety profile of LTP by recording the presence of adverse events such as bleeding, perforation, and infection in both initial and crossover phases from during the procedure up to 8 weeks post-procedure.
Clinical Improvement of Gastrointestinal Symptoms | Baseline, 8 Weeks
  Change in Gastrointestinal Symptoms from Baseline Using the gastrointestinal symptom rating scale (GSRS). This has a seven-point graded Likert-type scale where 1 represents absence of troublesome symptoms and 7 represents very troublesome symptoms.
Change in quality of life score from baseline using the 12 item Short Form Survey (SF-12) | Baseline, 8 Weeks
  Comparison of quality of life scores from baseline to 4 weeks post-treatment using the SF-12 scoring system. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning. A score of 50 or less has been recommended as a cut-off to determine a physical condition in the Physical Health Composite Score (PCS) section; while a score of 42 or less may be indicative of 'clinical depression' Mental Health Composite Score (MCS) section.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher C. Thompson, MD, MSc, Principal Investigator — Brigham and Womens Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual Participant Data (IPD) will be shared on a case by case basis with an Institutional data transfer agreement in place.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: 12 months after publication.
Access Criteria: IPD requests should be made directly to the PI who will determine feasibility of the request. Institutional data transfer agreement will need to be executed to share data.

REFERENCES:
- [Background] Angrisani L, Santonicola A, Iovino P, Ramos A, Shikora S, Kow L. Bariatric Surgery Survey 2018: Similarities and Disparities Among the 5 IFSO Chapters. Obes Surg. 2021 May;31(5):1937-1948. doi: 10.1007/s11695-020-05207-7. Epub 2021 Jan 12. PMID 33432483
- [Background] Sapala JA, Wood MH, Sapala MA, Flake TM Jr. Marginal ulcer after gastric bypass: a prospective 3-year study of 173 patients. Obes Surg. 1998 Oct;8(5):505-16. doi: 10.1381/096089298765554061. PMID 9819081
- [Background] Coblijn UK, Goucham AB, Lagarde SM, Kuiken SD, van Wagensveld BA. Development of ulcer disease after Roux-en-Y gastric bypass, incidence, risk factors, and patient presentation: a systematic review. Obes Surg. 2014 Feb;24(2):299-309. doi: 10.1007/s11695-013-1118-5. PMID 24234733
- [Background] Steinemann DC, Bueter M, Schiesser M, Amygdalos I, Clavien PA, Nocito A. Management of anastomotic ulcers after Roux-en-Y gastric bypass: results of an international survey. Obes Surg. 2014 May;24(5):741-6. doi: 10.1007/s11695-013-1152-3. PMID 24347350
- [Background] Choi J, Polistena C. Management of Marginal Ulceration. In: Camacho D, Zundel N, eds. Complications in Bariatric Surgery. Cham: Springer International Publishing; Imprint: Springer; 2018: 45-58
- [Background] Carr WR, Mahawar KK, Balupuri S, Small PK. An evidence-based algorithm for the management of marginal ulcers following Roux-en-Y gastric bypass. Obes Surg. 2014 Sep;24(9):1520-7. doi: 10.1007/s11695-014-1293-z. PMID 24851857
- [Background] Adamovich I, Agarwal S, Ahedo E et al. The 2022 Plasma Roadmap: low temperature plasma science and technology. Plasma Sources Sci. Technol. 2022; 55: 373001
- [Background] Chuangsuwanich A, Assadamongkol T, Boonyawan D. The Healing Effect of Low-Temperature Atmospheric-Pressure Plasma in Pressure Ulcer: A Randomized Controlled Trial. Int J Low Extrem Wounds. 2016 Dec;15(4):313-319. doi: 10.1177/1534734616665046. Epub 2016 Sep 20. PMID 27581113
- [Background] Mirpour S, Fathollah S, Mansouri P, Larijani B, Ghoranneviss M, Mohajeri Tehrani M, Amini MR. Cold atmospheric plasma as an effective method to treat diabetic foot ulcers: A randomized clinical trial. Sci Rep. 2020 Jun 26;10(1):10440. doi: 10.1038/s41598-020-67232-x. PMID 32591594
- [Background] Hartwig S, Preissner S, Voss JO, Hertel M, Doll C, Waluga R, Raguse JD. The feasibility of cold atmospheric plasma in the treatment of complicated wounds in cranio-maxillo-facial surgery. J Craniomaxillofac Surg. 2017 Oct;45(10):1724-1730. doi: 10.1016/j.jcms.2017.07.008. Epub 2017 Jul 27. PMID 28843407
- [Background] Isbary G, Morfill G, Schmidt HU, Georgi M, Ramrath K, Heinlin J, Karrer S, Landthaler M, Shimizu T, Steffes B, Bunk W, Monetti R, Zimmermann JL, Pompl R, Stolz W. A first prospective randomized controlled trial to decrease bacterial load using cold atmospheric argon plasma on chronic wounds in patients. Br J Dermatol. 2010 Jul;163(1):78-82. doi: 10.1111/j.1365-2133.2010.09744.x. Epub 2010 Mar 5. PMID 20222930
- [Background] Abu Rached N, Kley S, Storck M, Meyer T, Stucker M. Cold Plasma Therapy in Chronic Wounds-A Multicenter, Randomized Controlled Clinical Trial (Plasma on Chronic Wounds for Epidermal Regeneration Study): Preliminary Results. J Clin Med. 2023 Aug 4;12(15):5121. doi: 10.3390/jcm12155121. PMID 37568525
- [Background] Bekeschus S, von Woedtke T, Emmert S, Schmidt A. Medical gas plasma-stimulated wound healing: Evidence and mechanisms. Redox Biol. 2021 Oct;46:102116. doi: 10.1016/j.redox.2021.102116. Epub 2021 Aug 28. PMID 34474394
- [Background] Graves DB. The emerging role of reactive oxygen and nitrogen species in redox biology and some implications for plasma applications to medicine and biology. Plasma Sources Sci. Technol. 2012; 45: 263001
- [Background] Gao J, Wang L, Xia C, Yang X, Cao Z, Zheng L, Ko R, Shen C, Yang C, Cheng C. Cold atmospheric plasma promotes different types of superficial skin erosion wounds healing. Int Wound J. 2019 Oct;16(5):1103-1111. doi: 10.1111/iwj.13161. Epub 2019 Jun 17. PMID 31207094
- [Background] Amini MR, Sheikh Hosseini M, Fatollah S, Mirpour S, Ghoranneviss M, Larijani B, Mohajeri-Tehrani MR, Khorramizadeh MR. Beneficial effects of cold atmospheric plasma on inflammatory phase of diabetic foot ulcers; a randomized clinical trial. J Diabetes Metab Disord. 2020 Jul 14;19(2):895-905. doi: 10.1007/s40200-020-00577-2. eCollection 2020 Dec. PMID 33520811
- [Background] Pekshev AV, Shekhter AB, Vagapov AB, Sharapov NA, Vanin AF. Study of plasma-chemical NO-containing gas flow for treatment of wounds and inflammatory processes. Nitric Oxide. 2018 Feb 28;73:74-80. doi: 10.1016/j.niox.2017.06.002. Epub 2017 Jun 26. PMID 28602888
- [Background] Schmidt A, Woedtke TV, Stenzel J, Lindner T, Polei S, Vollmar B, Bekeschus S. One Year Follow-Up Risk Assessment in SKH-1 Mice and Wounds Treated with an Argon Plasma Jet. Int J Mol Sci. 2017 Apr 19;18(4):868. doi: 10.3390/ijms18040868. PMID 28422070
- [Background] Metelmann H-R, Vu TT, Do HT et al. Scar formation of laser skin lesions after cold atmospheric pressure plasma (CAP) treatment: A clinical long term observation. Clinical Plasma Medicine 2013; 1: 30-35
- [Background] Rutkowski R, Daeschlein G, von Woedtke T, Smeets R, Gosau M, Metelmann HR. Long-term Risk Assessment for Medical Application of Cold Atmospheric Pressure Plasma. Diagnostics (Basel). 2020 Apr 11;10(4):210. doi: 10.3390/diagnostics10040210. PMID 32290487
- [Background] Winter J, Brandenburg R, Weltmann K-D. Atmospheric pressure plasma jets: an overview of devices and new directions. Plasma Sources Sci. Technol. 2015; 24: 64001
- [Background] Grund KE, Zindel C, Farin G. [Argon plasma coagulation through a flexible endoscope. Evaluation of a new therapeutic method after 1606 uses]. Dtsch Med Wochenschr. 1997 Apr 4;122(14):432-8. doi: 10.1055/s-2008-1047634. German. PMID 9138921
- [Background] Zenker M. Argon plasma coagulation. GMS Krankenhhyg Interdiszip. 2008 Nov 3;3(1):Doc15. PMID 20204117
- [Background] Eickhoff A, Jakobs R, Schilling D, Hartmann D, Weickert U, Enderle MD, Eickhoff JC, Riemann JF. Prospective nonrandomized comparison of two modes of argon beamer (APC) tumor desobstruction: effectiveness of the new pulsed APC versus forced APC. Endoscopy. 2007 Jul;39(7):637-42. doi: 10.1055/s-2007-966571. PMID 17611919
- [Background] Kwan V, Bourke MJ, Williams SJ, Gillespie PE, Murray MA, Kaffes AJ, Henriquez MS, Chan RO. Argon plasma coagulation in the management of symptomatic gastrointestinal vascular lesions: experience in 100 consecutive patients with long-term follow-up. Am J Gastroenterol. 2006 Jan;101(1):58-63. doi: 10.1111/j.1572-0241.2006.00370.x. PMID 16405534
- [Background] Vargo JJ. Clinical applications of the argon plasma coagulator. Gastrointest Endosc. 2004 Jan;59(1):81-8. doi: 10.1016/s0016-5107(03)02296-x. No abstract available. PMID 14722558
- [Background] Grund KE, Straub T, Farin G. New haemostatic techniques: argon plasma coagulation. Baillieres Best Pract Res Clin Gastroenterol. 1999 Apr;13(1):67-84. doi: 10.1053/bega.1999.0009. PMID 11030635
- [Background] Grund KE, Storek D, Farin G. Endoscopic argon plasma coagulation (APC) first clinical experiences in flexible endoscopy. Endosc Surg Allied Technol. 1994 Feb;2(1):42-6. PMID 8081915
- [Background] Weiss M, Utz R, Ackermann M et al. Characterization of a non-thermally operated electrosurgical argon plasma source by electron spin resonance spectroscopy. Plasma Process Polym 2019; 16: 1800150
- [Background] Weiss M, Arnholdt M, Hissnauer A, Fischer I, Schonfisch B, Andress J, Gerstner S, Dannehl D, Bosmuller H, Staebler A, Brucker SY, Henes M. Tissue-preserving treatment with non-invasive physical plasma of cervical intraepithelial neoplasia-a prospective controlled clinical trial. Front Med (Lausanne). 2023 Aug 15;10:1242732. doi: 10.3389/fmed.2023.1242732. eCollection 2023. PMID 37654659